CLINICAL TRIAL: NCT05998161
Title: Evaluating the Effectiveness of a Digital Therapeutic (Reviga) for People With Stress or Burnout - a Randomized Controlled Trial
Brief Title: Evaluating the Effectiveness of a Digital Therapeutic (Reviga) for People With Stress or Burnout
Acronym: LAVENDER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gaia AG (Industry)
Collaborators: University Hospital Schleswig-Holstein (Other); Hannover Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: reviga RCT 2023
Record Dates: First submitted 2023-08-09; First posted 2023-08-18 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Stress; Burnout
MeSH Terms: conditions — Burnout, Psychological

STUDY DESIGN:
Masking Description: All endpoints are patient-reported outcome measures (PROMs). Given that participants are aware of their study group (receiving reviga in addition to treatment as usual or only receiving treatment as usual), this trial is not blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- reviga + TAU (Experimental): Participants allocated to the intervention group will receive access to reviga in addition to treatment as usual (TAU).
  reviga is a digital health application designed for individuals with stress and burnout, accessible through a web browser. The application focuses on treatment methods derived from cognitive behavioral therapy (CBT). Topics addressed by reviga are relaxation, psychoeducation and exercises regarding relevant cognitions and behavior, acceptance, relationships, problem solving strategies, and positive psychology.
  The program operates through interactive "dialogues", which are accompanied by illustrations, audio recordings, motivating text messages, worksheets, and summaries. Users are also encouraged to regularly complete short questionnaires to monitor their complaints. Once registered, the program remains accessible for 180 days.
  Interventions: Behavioral: reviga
- TAU (No Intervention): Participants allocated to the control group will receive access to treatment as usual (TAU).

INTERVENTIONS:
Behavioral: reviga — Participants will receive access to the digital health intervention reviga in addition to TAU.
  Arms: reviga + TAU

SUMMARY:
In this single-blinded randomized controlled clinical trial 290 patients with stress or burnout will be investigated regarding the effectiveness of a digital therapeutic for improvement of stress level, the unguided online intervention reviga.

Inclusion criteria are: age 18-65 years, ICD-10 diagnosis Z73, operationalized as above average general stress level (PSS score > 21) and increased levels of work-related stress / burnout (OLBI score ≥ 2.18), living in Germany, working a minimum of 20h per week, having a stable treatment for at least 30 days at the time of inclusion, and consent to participation. Exclusion criterion is having plans to change the treatment in the upcoming three months at the time of inclusion.

Patients will be randomized and allocated to either an intervention group, receiving reviga in addition to treatment as usual (TAU), or a control group, receiving only TAU. The control group will be granted access to the program at the end of the study. Primary endpoint will be the perceived stress measured by the PSS score, with three months post-allocation being the primary time point for assessment of effectiveness. Six months post allocation will be used as a timepoint for follow-up assessment of endpoints. Secondary endpoints will be anxiety symptoms, level of functioning, burnout symptoms, health-related quality of life, and sick days.

ELIGIBILITY:
Inclusion Criteria:

* age 18-65 years
* living in Germany
* employed (minimum of 20h/week)
* ICD-10 diagnosis Z73, operationalized as above average general stress level (PSS score > 21) and increased levels of work-related stress / burnout (OLBI score ≥ 2.18)
* stable treatment (psychotherapy, medication, no treatment) for at least 30 days at the time of inclusion
* consent to participation

Exclusion Criteria:

* plans to change treatment (psychotherapy, medication, ...) in the upcoming three months at the time of inclusion

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 290 (Actual)
Dates: Start 2023-09-04 (Actual); Primary Completion 2024-06-22 (Actual); Study Completion 2024-06-22 (Actual)

PRIMARY OUTCOMES:
Stress symptoms | 3 months
  Perceived Stress Scale (PSS-10). Total score ranging from 0-40; higher scores mean more stress symptoms (worse outcome).

SECONDARY OUTCOMES:
Anxiety symptoms | 3 months, 6 months
  Generalized Anxiety Assessment (GAD-7). Total score ranging from 0-21; higher scores mean higher anxiety (worse outcome).
Functioning | 3 months, 6 months
  Work and Social Adjustment Scale (WSAS). Total score ranging from 0-40; higher scores mean higher impairment (worse outcome).
Burnout symptoms | 3 months, 6 months
  Oldenburg Burnout Inventory (OLBI). Two subscales (exhaustion and disengagement), each ranging from 8-32; higher scores mean higher burnout symptoms (worse outcome).
Health-related quality of life | 3 months, 6 months
  Assessment of Quality of Life - 8D (AQoL-8D). AQoL-8D score ranging from 0-100; higher scores mean higher quality of life (better outcome).
Sick days | 3 months, 6 months
  Number of sick days in the past 3 months
Stress symptoms | 6 months
  Perceived Stress Scale (PSS-10). Total score ranging from 0-40; higher scores mean more stress symptoms (worse outcome).

OTHER OUTCOMES:
Depressive symptoms | 3 months, 6 months
  Patient Health Questionnaire - 9 item version (PHQ-9). Total score ranging from 0-27; higher scores mean higher depressive symptoms (worse outcome).
Effort and reward imbalance | 3 months, 6 months
  Effort-reward-imbalance (ERI). Three subscales: effort, ranging from 3-12, higher scores mean higher effort; reward, ranging from 7=28, higher scores mean higher reward; over-commitment, ranging from 6-24, higher scores mean higher over-commitment. Ratio effort/reward: scores >1 mean more efforts for each reward (worse outcome).
hospital stays | 3 months, 6 months
  Number of hospital stays in the past 3 months
curative stays | 3 months, 6 months
  Number of curative stays in the past 3 months
doctor visits | 3 months, 6 months
  Number of doctor visits in the past 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Kamila Jauch-Chara, MD, Principal Investigator — Universitätsklinikum Schleswig-Holstein, Campus Kiel, Klinik für Psychosomatik und Psychotherapie, Zentrum für Integrative Psychiatrie, Michaelistraße 1, 24105 Kiel
Locations (1):
- GAIA AG, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No